CLINICAL TRIAL: NCT06197841
Title: Neurofilament Light Chain and Cognitive Impairment as Diagnostic and Prognostic Markers in naïve Multiple Sclerosis Patients
Brief Title: Neurofilament Light Chain as Diagnostic and Prognostic Marker in naïve Multiple Sclerosis Patients
Acronym: NFLMS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, professor of Neurology, Assiut University
Other Study IDs: Assiut University/Egypt
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Role of Neurofilment in Diagnosis of Multiple Sclerosis
Keywords: Naïve multiple sclerosis patients; cognitive impairment; Neurofilment light chain; Chitinase; diagnosis and predictor for outcome
MeSH Terms: conditions — Cognitive Dysfunction; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neurofilament protein detected in the serum appears to be a good marker for the extent of active neurodegeneration. Chitinase may also be a good marker reflecting the degree of astrocyte activation, or damage in active lesions (Paul et al, 2018).These markers have some clinical value for diagnosis and monitoring of disease activity. NfL can be objectively measured and quantified, it is highly sensitive to neurodegenerative processes and its concentration changes as the disease worsens or improves (Disanto et al., 2017). Numerous studies have shown that NfL levels increase during MS relapses and correlate with MRI lesion development (Disanto et al., 2016, 2017; Novakova et al., 2017), disease activity, (Thebault et al., 2020). Cognitive impairment is common in the early stages of multiple sclerosis, mainly affecting attention, working memory, and information processing speed, but also memory, inhibition, and conceptualisation. Poor performance is common but remains subtle and does not significantly affect the quality of life at this stage. However, many studies shows that these deficits reflect the destruction both within and outside lesions, and that they may therefore be considered as a severity marker in the early stages of multiple sclerosis. (Lengenfelder et al., 2005).

The aim of the work is to detect the role of serum NFL and chitinase as biomarkers in the diagnosis and prognosis of newly diagnosed multiple sclerosis patients, and to estimate the incidence of cognitive impairment and their relationship with the NFL in newly diagnosed MS patients.

DETAILED DESCRIPTION:
Many immunological studies have been performed with the aim to identify MS specific biomarkers and disease mechanisms and to find markers able to predict clinical disease course and outcome (Housley et al, 2015) Besides MRI and markers related to therapy (induction of blocking antibodies) or JC virus infection, they include markers for neurodegeneration, such as neurofilaments, markers for astrocytic activation (eg. chitinase or GFAP). Neurofilament protein detected in the serum or cerebrospinal fluid appears to be a good marker for the extent of active neurodegeneration, but this is not MS specific. Chitinase may be a good marker for active disease in RRMS, reflecting the degree of astrocyte activation, or damage in active lesions (Paul et al, 2018).These markers have some clinical value for diagnosis and monitoring of disease activity. Cognitive impairment is common in the early stages of multiple sclerosis, mainly affecting attention, working memory, and information processing speed, but also memory, inhibition, and conceptualisation. Poor performance is common but remains subtle and does not significantly affect the quality of life at this stage. However, many studies shows that these deficits reflect the destruction both within and outside lesions, and that they may therefore be considered as a severity marker in the early stages of multiple sclerosis. (Lengenfelder et al., 2005).Aim of the work The aim of the work is to detect the role of serum neurofilament light chain and chitinase as well as cognitive impairment as biomarkers in the diagnosis and prognosis of newly diagnosed multiple sclerosis patients, and to estimate the incidence of cognitive impairment and their relationship with the NFL in newly diagnosed MS patients.Study Design This study is a cross-sectional, prospective, observational study. Subjects All newly diagnosed cases With MS patients attending different MS unites in Assiut governorate will be recruited and all eligible patients will be included.

Inclusion criteria:

All patients newly diagnosed MS according to the 2017-McDonalds criteria.

Exclusion criteria:

1. patients who are already diagnosed as MS and on treatment.
2. Presence of other disorder or on medications that may affect the neurological or cognitive disorders.
3. Patients failed to commit to the follow up visits and regular MRI scans
4. Patients refused to sign the written informed consent

Patients who will meet the inclusion and exclusion criteria will be assessed in the 1st visit by direct interview followed by clinical examination and neuropsychological assessments as well as laboratory assessment. Baseline MRI scans will be obtained at the first visit and 12 months. In the follow up visits every 6 months for 1and half year at least with assessment for all previous will be repeated to detect early signs of progression.Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

Demographic data: age at presentation and age at onset, sex, education years and special habits Clinical data: duration of illness, until diagnosis number of relapses/year and their features.

Clinical assessment: EDSS, 9-hole pig test, 25-feet walking test.

Clinical rating scales :

Cognitive assessment using the Brief International Cognitive Assessment for Multiple sclerosis (BICAMS) with the Arabic validated version (8) that include:

Symbol Digit Modalities Test (SDMT) (Langdon et al. 2012) for evaluating the information processing speed.

California Verbal Learning Test (CVLT-II) for evaluating verbal learning and memory.

Brief Visual Memory Test (BVMT) for evaluating visual learning and memory.

Multiple sclerosis Quality of life MSQoL-54 questionnaire (10) with sub scales that measures physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function.

Hamilton depression rating-17-item version (HAM-D 17).

Laboratory investigation:

CSF Oligoclonal band, Serum light chain Neurofilament using PCR Research outcomes The primary outcome is the detection of neurofilament as diagnostic and prognostic inflammatory markers in newly diagnosed MS patients.

Secondary outcome measure is incidence of depression, cognitive impairment in newly diagnosed MS patients.

Follow up of each patient every 6 months using the same previous scales

ELIGIBILITY:
Inclusion Criteria:

All patients newly diagnosed MS according to the 2017-McDonalds criteria.

Exclusion criteria:

1. patients who are already diagnosed MS and under DMTs treatment
2. Presence of other disorder or on medications that may affect the neurological or cognitive disorders.
3. Patients failed to commit to the follow up visits and regular MRI scans
4. Patients refused to sign the written informed consent

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Naïve Patients who will meet the inclusion and exclusion criteria of MS will be assessed in the 1st visit by direct interview followed by clinical examination and neuropsychological assessments as well as laboratory assessment. Baseline MRI scans will be obtained at the first visit and 12, months follow up. In the follow up visits every 6 months for 1and half year at least with assessment for all previous will be repeated to detect early signs of progression.
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the detection of neurofilament light chain as diagnostic and prognostic inflammatory markers in newly diagnosed MS patients. | 1 and half year
  Assessment of the serum level of NFL at base line before starting DMT and correlate it with motor disability, cognitive impairment after one and half year

SECONDARY OUTCOMES:
Assessment of the incidence of cognitive impairment among naive multiple sclerosis patients and their correlation with neurofilment light chain | 1 and half year
  Assessment of cognitive impairment of the MS Patients using BICAMS

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed El menshawy, Asyut, Egypt

REFERENCES:
- [Derived] Khedr EM, Hassan MM, Ezzeldeen MY, El-Kady MS, El-Mokhtar MA, Shokry AE. Motor symptoms at onset and manual dexterity predict cognitive impairment in drug-naive individuals with multiple sclerosis. J Neuroimmunol. 2025 Apr 15;401:578571. doi: 10.1016/j.jneuroim.2025.578571. Epub 2025 Feb 25. PMID 40022906